CLINICAL TRIAL: NCT05225727
Title: Me & You-Tech: A Socio-Ecological Solution to Teen Dating Violence for the Digital Age
Acronym: MYTech
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Radiant Creative Group, LLC (Industry); University of Texas (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Melissa Peskin, Professor, Department of Health Promotion and Behavioral Sciences, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSC-SPH-19-0253; R42HD100233-01 (NIH)
Record Dates: First submitted 2022-01-24; First posted 2022-02-04 (Actual); Results first posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Adolescent Behavior; Interpersonal Relations; Domestic Violence; Physical Violence
Keywords: adolescent behavior; interpersonal relationships; intimate partner violence; Violence/prevention & control; program evaluation; teen dating violence; programs using technology
MeSH Terms: conditions — Adolescent Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Students randomized to the intervention group will receive Me & You Tech in place of their standard health education.
  Interventions: Behavioral: Me & You - Tech
- Control (No Intervention): Students assigned to the standard care condition will receive their usual health education which usually includes knowledge-based content on violence prevention taught from the state textbook

INTERVENTIONS:
Behavioral: Me & You - Tech — The 13 MYT lessons will train youth to adopt a zero tolerance approach to dating violence (DV) and contain activities to enable youth to recognize healthy (non-abusive) and unhealthy (abusive) relationships, assess their own relationships, and adopt and practice a lifestyle paradigm of select-detect-protect informed by SCT self-regulatory frameworks. Within this lifestyle paradigm, youth select their personal rules to have only healthy (non-abusive) relationships, detect unhealthy (abusive) relationships that might threaten their rules, and learn to protect their rules using communication, management, and avoidance skills. MYT will tailor content by gender, relationship status, and the youth's DV profile of perpetration or victimization based on the Conflict in Adolescent Dating and Relationship Inventory (CADRI).
  Arms: Intervention

SUMMARY:
The purpose of this study is to develop and evaluate a multi-level (youth, parent, school) Internet-based dating violence prevention program, 'Me & You-Tech' (MYT) for 6th-grade middle school students.

DETAILED DESCRIPTION:
The purpose of this three year study is to develop and evaluate Me & You - Tech, a computer-based healthy relationships and dating violence prevention curriculum for 6th grade students. The curriculum will be developed and adapted from an existing effective healthy relationship curriculum, Me & You: Building Healthy Relationships. A randomized two-arm design will be conducted among 6th grade students, where students receiving the curriculum were compared to students receiving usual care. Four middle schools participated in the study, 2 schools were randomly assigned to receive the curriculum and two to receive usual care. Outcomes were assessed at baseline, 3 months following completion of the intervention, and 9 months after baseline. Parental permission and student assent were obtained prior to administration of the surveys. The primary hypothesis is that students who receive the curriculum will have significantly lower teen dating violence perpetration than those who do not receive the curriculum.

ELIGIBILITY:
Inclusion Criteria:

* 6th grade student
* Currently attending a middle school

Exclusion Criteria:

* Previous participation in usability and feasibility testing
* Inability to complete activities
* Inability to read English
* Lack of home internet connectivity

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 123 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-12-14 (Actual); Study Completion 2024-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Peskin, PhD, Principal Investigator — University of Texas Houston School of Public Health; Ross Shegog, PhD, Principal Investigator — University of Texas Houston School of Public Health
Locations (1):
- University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Schools
Period: Overall Study
Arm/Group | Intervention | Control
Started | 43; 2 Schools | 80; 2 Schools
Follow up 1 (about 2 months after baseline) | 26; 2 Schools | 58; 2 Schools
Follow up 2 (6 months after baseline) | 30; 2 Schools | 49; 2 Schools
Completed | 30; 2 Schools | 49; 2 Schools
Not Completed | 13; 0 Schools | 31; 0 Schools

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 43 | 80 | 123
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Data were not collected from 1 participant in the control arm because they did not answer this question.
  years
    number analyzed (Participants) | 43 | 79 | 122
    (all) | 11.8 (0.72) | 11.8 (0.67) | 11.8 (0.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 43 | 62
  Male | 24 | 37 | 61
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 22 | 44 | 66
  Black/African American | 15 | 25 | 40
  Other | 5 | 10 | 15
  Unknown | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 43 | 80 | 123

OUTCOME MEASURES:

1. Primary Outcome: Number of Youth Who Perpetrated Any Type of Teen Dating Violence as Assessed by the Conflict in Adolescent Dating Relationships Inventory (CADRI)
Description: The CADRI is a 34-item questionnaire that assesses abusive behavior among adolescent dating partners (Wolfe et al., 2001). The scale has a count score ranging from 0-34. If the score is 1 or more, teen dating violence perpetration occurred. Those in the Category of "Yes" have a score of 1 or more and are considered perpetrators. Those in the Category of "No" have a score of 0 and either did not report a dating partner or reported a dating partner but did not report perpetration.
Time Frame: Baseline
Population: Data were not collected from 5 participants in the Intervention arm because they did not complete the question. Data were not collected from 6 participants in the Control arm because they did not complete the question
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 38 | 74
Participants
  "Yes" Considered Perpetrators | 12 | 15
  "No" Not Considered Perpetrators | 26 | 59

2. Primary Outcome: Number of Youth Who Perpetrated Any Type of Teen Dating Violence as Assessed by the Conflict in Adolescent Dating Relationships Inventory (CADRI)
Description: as for outcome 1
Time Frame: 6 months after baseline
Population: Data were not collected from 4 participants in the Intervention arm because they did not complete the question. Data were not collected from 3 participants in the Control arm because they did not complete the question.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 26 | 46
Participants
  "Yes" Considered Perpetrators | 4 | 9
  "No" Not Considered Perpetrators | 22 | 37

3. Primary Outcome: Number of Youth Who Were Victimized by Any Type of Teen Dating Violence as Assessed by the Conflict in Adolescent Dating Relationships Inventory (CADRI)
Description: The CADRI is a 34-item questionnaire that assesses abusive behavior among adolescent dating partners (Wolfe et al., 2001). The scale has a count score ranging from 0-34. If the score is 1 or more, teen dating violence victimization occurred. Those in the Category of "Yes" have a score of 1 or more and are considered victims. Those in the Category of "No" have a score of 0 and either did not report a dating partner or reported a dating partner but did not report victimization.
Time Frame: Baseline
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 38 | 74
Participants
  "Yes" Considered Victims | 10 | 18
  "No" Not Considered Victims | 28 | 56

4. Primary Outcome: Number of Youth Who Were Victimized by Any Type of Teen Dating Violence as Assessed by the Conflict in Adolescent Dating Relationships Inventory (CADRI)
Description: as for outcome 3
Time Frame: 6 months after baseline
Population: Data were not collected from 4 participants in the Intervention arm because they did not complete the question. Data were not collected from 4 participants in the Control arm because they did not complete the question.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 26 | 45
Participants
  "Yes" Considered Victims | 3 | 5
  "No" Not Considered Victims | 23 | 40

5. Secondary Outcome: Number of Youth Who Perpetrated Psychological Teen Dating Violence as Assessed by the Conflict in Adolescent Dating Relationships Inventory (CADRI) - Psychological Perpetration Subscale
Description: The CADRI is a 34-item questionnaire that assesses abusive behavior among adolescent dating partners (Wolfe et al., 2001). It includes a 13-item psychological perpetration subscale with a count score ranging from 0-13. If the score is 3 or more, psychological perpetration occurred. Those in the Category of "Yes" have a score of 3 or more and are considered perpetrators. Those in the Category of "No" have a score of 0, 1, or 2 and either did not report a dating partner or reported a dating partner but did not report psychological perpetration.
Time Frame: Baseline
Population: Data were not collected from 5 participants in the Intervention arm because they did not complete the question. Data were not collected from 4 participants in the Control arm because they did not complete the question.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 38 | 76
Participants
  "Yes" Considered Perpetrators | 6 | 9
  "No" Not Considered Perpetrators | 32 | 67

6. Secondary Outcome: Number of Youth Who Perpetrated Psychological Teen Dating Violence as Assessed by the Conflict in Adolescent Dating Relationships Inventory (CADRI) - Psychological Perpetration Subscale
Description: as for outcome 5
Time Frame: 6 months after baseline
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 26 | 46
Participants
  "Yes" Considered Perpetrators | 1 | 4
  "No" Not Considered Perpetrators | 25 | 42

7. Secondary Outcome: Number of Youth Who Were Victimized by Psychological Teen Dating Violence as Assessed by the Conflict in Adolescent Dating Relationships Inventory (CADRI) - Psychological Victimization Subscale
Description: The CADRI is a 34-item questionnaire that assesses abusive behavior among adolescent dating partners (Wolfe et al., 2001). It includes a 13-item psychological victimization subscale with a count score ranging from 0-13. If the score is 3 or more, psychological victimization occurred. Those in the Category of "Yes" have a score of 3 or more and are considered victims. Those in the Category of "No" have a score of 0, 1, or 2 and either did not report a dating partner or reported a dating partner but did not report psychological victimization.
Time Frame: Baseline
Population: Data were not collected from 5 participants in the Intervention arm because they did not complete the question. Data were not collected from 5 participants in the Control arm because they did not complete the question.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 38 | 75
Participants
  "Yes" Considered Victims | 7 | 12
  "No" Not Considered Victims | 31 | 63

8. Secondary Outcome: Number of Youth Who Were Victimized by Psychological Teen Dating Violence as Assessed by the Conflict in Adolescent Dating Relationships Inventory (CADRI) - Psychological Victimization Subscale
Description: as for outcome 7
Time Frame: 6 months after baseline
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 26 | 45
Participants
  "Yes" Considered Victims | 2 | 5
  "No" Not Considered Victims | 24 | 40

9. Secondary Outcome: Number of Youth Who Perpetrated Physical Teen Dating Violence as Assessed by the Conflict in Adolescent Dating Relationships Inventory (CADRI) - Physical Perpetration Subscale
Description: The CADRI is a 34-item questionnaire that assesses abusive behavior among adolescent dating partners (Wolfe et al., 2001). It includes a 4-item physical perpetration subscale with a count score ranging from 0-4. If the score is 1 or more, physical perpetration occurred. Those in the Category of "Yes" have a score of 1 or more and are considered perpetrators. Those in the Category of "No" have a score of 0 and either did not report a dating partner or reported a dating partner but did not report physical perpetration.
Time Frame: Baseline
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 38 | 76
Participants
  "Yes" Considered Perpetrators | 4 | 9
  "No" Not Considered Perpetrators | 34 | 67

10. Secondary Outcome: Number of Youth Who Perpetrated Physical Teen Dating Violence as Assessed by the Conflict in Adolescent Dating Relationships Inventory (CADRI) - Physical Perpetration Subscale
Description: as for outcome 9
Time Frame: 6 months after baseline
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 26 | 46
Participants
  "Yes" Considered Perpetrators | 1 | 4
  "No" Not Considered Perpetrators | 25 | 42

11. Secondary Outcome: Number of Youth Who Were Victimized by Physical Teen Dating Violence as Assessed by the Conflict in Adolescent Dating Relationships Inventory (CADRI) - Physical Victimization Subscale
Description: The CADRI is a 34-item questionnaire that assesses abusive behavior among adolescent dating partners (Wolfe et al., 2001). It includes a 4-item physical victimization subscale with a count score ranging from 0-4. If the score is 1 or more, physical victimization occurred. Those in the Category of "Yes" have a score of 1 or more and are considered victims. Those in the Category of "No" have a score of 0 and either did not report a dating partner or reported a dating partner but did not report physical victimization.
Time Frame: Baseline
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 38 | 75
Participants
  "Yes" Considered Victims | 6 | 10
  "No" Not Considered Victims | 32 | 65

12. Secondary Outcome: Number of Youth Who Were Victimized by Physical Teen Dating Violence as Assessed by the Conflict in Adolescent Dating Relationships Inventory (CADRI) - Physical Victimization Subscale
Description: as for outcome 11
Time Frame: 6 months after baseline
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 26 | 45
Participants
  "Yes" Considered Victims | 0 | 3
  "No" Not Considered Victims | 26 | 42

13. Secondary Outcome: Number of Youth Who Perpetrated Sexual Teen Dating Violence as Assessed by the Conflict in Adolescent Dating Relationships Inventory (CADRI) - Sexual Perpetration Subscale
Description: The CADRI is a 34-item questionnaire that assesses abusive behavior among adolescent dating partners (Wolfe et al., 2001). One sexual perpetration item was used with a count score ranging from 0-1. If the score is 1, sexual perpetration occurred. Those in the Category of "Yes" have a score of 1 and are considered perpetrators. Those in the Category of "No" have a score of 0 and either did not report a dating partner or reported a dating partner but did not report sexual perpetration.
Time Frame: Baseline
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 38 | 74
Participants
  "Yes" Considered Perpetrators | 0 | 3
  "No" Not Considered Perpetrators | 38 | 71

14. Secondary Outcome: Number of Youth Who Perpetrated Sexual Teen Dating Violence as Assessed by the Conflict in Adolescent Dating Relationships Inventory (CADRI) - Sexual Perpetration Subscale
Description: as for outcome 13
Time Frame: 6 months after baseline
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 26 | 46
Participants
  "Yes" Considered Perpetrators | 0 | 0
  "No" Not Considered Perpetrators | 26 | 46

15. Secondary Outcome: Number of Youth Who Were Victimized by Sexual Teen Dating Violence as Assessed by the Conflict in Adolescent Dating Relationships Inventory (CADRI) - Sexual Victimization Subscale
Description: The CADRI is a 34-item questionnaire that assesses abusive behavior among adolescent dating partners (Wolfe et al., 2001). One sexual victimization item was used with a count score ranging from 0-1. If the score is 1, sexual victimization occurred. Those in the Category of "Yes" have a score of 1 and are considered victims. Those in the Category of "No" have a score of 0 and either did not report a dating partner or reported a dating partner but did not report sexual victimization.
Time Frame: Baseline
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 38 | 74
Participants
  "Yes" Considered Victims | 2 | 6
  "No" Not Considered Victims | 36 | 68

16. Secondary Outcome: Number of Youth Who Were Victimized by Sexual Teen Dating Violence as Assessed by the Conflict in Adolescent Dating Relationships Inventory (CADRI) - Sexual Victimization Subscale
Description: as for outcome 15
Time Frame: 6 months after baseline
Population: Data were not collected from 4 participants in the Intervention arm because they did not complete the question. Data were not collected from 4 participants in the Control arm they did not complete the question.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 26 | 45
Participants
  "Yes" Considered Victims | 0 | 1
  "No" Not Considered Victims | 26 | 44

17. Secondary Outcome: Number of Youth Who Perpetrated Digital Teen Dating Violence as Assessed by a Cyber Dating Abuse Questionnaire - Perpetrator Subscale
Description: The Cyber Dating Abuse questionnaire include 22 questions relating to cyber dating abuse among dating partners adapted from existing sources (Zweig et al., 2014; Picard, 2007). It includes a 12-item cyber dating abuse perpetration subscale with a count score ranging from 0-11. If the score is 1 or more, cyber abuse perpetration occurred. Those in the Category of "Yes" have a score of 1 and are considered perpetrators. Those in the Category of "No" have a score of 0 and either did not report a dating partner or reported a dating partner but did not report cyber perpetration.
Time Frame: Baseline
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 38 | 75
Participants
  "Yes" Considered Perpetrators | 9 | 12
  "No" Not Considered Perpetrators | 29 | 63

18. Secondary Outcome: Number of Youth Who Perpetrated Digital Teen Dating Violence as Assessed by the Cyber Dating Abuse Questionnaire - Perpetrator Subscale
Description: as for outcome 17
Time Frame: 6 months after baseline
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 26 | 45
Participants
  "Yes" Considered Perpetrators | 4 | 8
  "No" Not Considered Perpetrators | 22 | 37

19. Secondary Outcome: Number of Youth Who Were Victimized by Digital Teen Dating Violence as Assessed by the Cyber Dating Abuse Questionnaire - Victimization Subscale
Description: The Cyber Dating Abuse questionnaire include 22 questions relating to cyber dating abuse among dating partners adapted from existing sources (Zweig et al., 2014; Picard, 2007). It includes a 12-item cyber dating abuse victimization subscale with a count score ranging from 0-11. If the score is 1 or more, cyber abuse victimization occurred. Those in the Category of "Yes" have a score of 1 and are considered victims. Those in the Category of "No" have a score of 0 and either did not report a dating partner or reported a dating partner but did not report cyber victimization.
Time Frame: Baseline
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 38 | 75
Participants
  "Yes" Considered Victims | 4 | 12
  "No" Not Considered Victims | 34 | 63

20. Secondary Outcome: Number of Youth Who Were Victimized by Digital Teen Dating Violence as Assessed by the Cyber Dating Abuse Questionnaire - Victimization Subscale
Description: The Cyber Dating Abuse questionnaire include 22 questions relating to cyber dating abuse among dating partners adapted from existing sources (Zweig et al., 2014; Picard, 2007). It includes a 12-item cyber dating abuse victimization subscale with a total score ranging from 0-11. If the score is 1 or more, cyber abuse victimization occurred. Those in the Category of "No" have a score of 0 and either did not report a dating partner or reported a dating partner but did not report cyber victimization.
Time Frame: 6 months after baseline
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 26 | 45
Participants
  "Yes" Considered Victims | 1 | 3
  "No" Not Considered Victims | 25 | 42

21. Secondary Outcome: Number of Youth Who Perpetrated Threatening Teen Dating Violence as Assessed by the Conflict in Adolescent Dating Relationships Inventory (CADRI) - Threatening Perpetration Subscale
Description: The CADRI is a 34-item questionnaire that assesses abusive behavior among adolescent dating partners (Wolfe et al., 2001). It includes a 4-item threatening perpetration subscale with a count score ranging from 0-4. If the score is 1 or more, threatening perpetration occurred. Those in the Category of "Yes" have a score of 1 or more and are considered perpetrators. Those in the Category of "No" have a score of 0 and either did not report a dating partner or reported a dating partner but did not report threatening perpetration.
Time Frame: Baseline
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 38 | 75
Participants
  "Yes" Considered Perpetrators | 1 | 2
  "No" Not Considered Perpetrators | 37 | 73

22. Secondary Outcome: Number Youth Who Perpetrated Threatening Teen Dating Violence as Assessed by the Conflict in Adolescent Dating Relationships Inventory (CADRI) - Threatening Perpetration Subscale
Description: as for outcome 21
Time Frame: 6 months after baseline
Population: Data were not collected from 4 participants in the Intervention arm they did not complete the question. Data were not collected from 3 participants in the Control arm because they did not complete the question.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 26 | 46
Participants
  "Yes" Considered Perpetrators | 0 | 3
  "No" Not Considered Perpetrators | 26 | 43

23. Secondary Outcome: Number of Youth Who Were Victimized by Threatening Teen Dating Violence as Assessed by the Conflict in Adolescent Dating Relationships Inventory (CADRI) - Threatening Victimization Subscale
Description: The CADRI is a 34-item questionnaire that assesses abusive behavior among adolescent dating partners (Wolfe et al., 2001). It includes a 4-item threatening victimization subscale with a count score ranging from 0-4. If the score is 1 or more, threatening victimization occurred. Those in the Category of "Yes" have a score of 1 or more and are considered victims. Reported are the participants with a score of 1 or more and 0. Those in the Category of "No" have a score of 0 and either did not report a dating partner or reported a dating partner but did not report threatening victimization.
Time Frame: Baseline
Population: Data were not collected from 5 participants in the Intervention arm because they did not complete the survey. Data were not collected from 6 participants in the Control arm because they did not complete the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 38 | 74
Participants
  "Yes" Considered Victims | 3 | 8
  "No" Not Considered Victims | 35 | 66

24. Secondary Outcome: Number of Youth Who Were Victimized by Threatening Teen Dating Violence as Assessed by the Conflict in Adolescent Dating Relationships Inventory (CADRI) - Threatening Victimization Subscale
Description: as for outcome 23
Time Frame: 6 months after baseline
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 26 | 45
Participants
  "Yes" Considered Victims | 1 | 2
  "No" Not Considered Victims | 25 | 43

25. Secondary Outcome: Student Norms Toward Violence as Assessed by the Acceptance of Dating Abuse Survey - Boys Aggressing Girls Subscale
Description: The Acceptance of Dating Abuse Survey is a questionnaire that assesses adolescents' perceptions of their norms toward violence for boys and girls (Foshee et al., 2001). A 6-item boys aggressing girls subscale is scored as 1 (Strongly Disagree) to 4 (Strongly Agree) for each item with a total average score ranging from 1-4. The higher the number, the more accepting of boys aggressing girls under certain circumstances.
Time Frame: Baseline
Population: Data were not collected from 3 participants in the Intervention arm because they did not answer this question. Data were not collected from 6 participants in the Control arm because they did not answer this question.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 40 | 74
score on a scale | 1.41 (0.53) | 1.46 (0.64)

26. Secondary Outcome: Student Norms Toward Violence as Assessed by the Acceptance of Dating Abuse Survey - Boys Aggressing Girls Subscale
Description: as for outcome 25
Time Frame: about 2 months after intervention
Population: Data were not collected from 1 participant in the Intervention arm because they did not answer this question. Data were not collected from 2 participants in the Control arm because they did not answer this question
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 25 | 56
score on a scale | 1.49 (0.62) | 1.41 (0.57)

27. Secondary Outcome: Student Norms Toward Violence as Assessed by the Acceptance of Dating Abuse Survey - Boys Aggressing Girls Subscale
Description: as for outcome 25
Time Frame: 6 months after intervention
Population: Data were not collected from 5 participants in the Intervention arm because they did not answer this question. Data were not collected from 1 participant in the Control arm because they did not answer this question.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 25 | 48
score on a scale | 1.68 (0.88) | 1.41 (0.60)

28. Secondary Outcome: Student Norms Toward Violence as Assessed by the Acceptance of Dating Abuse Survey- Girls Aggressing Boys Subscale
Description: The Acceptance of Dating Abuse Survey is a questionnaire that assesses adolescents' perceptions of their norms toward violence for boys and girls (Foshee et al., 2001). A 4-item girls aggressing boys subscale is scored as 1 (Strongly Disagree) to 4 (Strongly Agree) for each item with a total average score ranging from 1-4. The higher the number, the more accepting of girls aggressing boys under certain circumstances.
Time Frame: Baseline
Population: Data were not collected from 4 participants in the Intervention arm because they did not answer this question. Data were not collected from 4 participants in the Control arm because they did not answer this question.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 39 | 76
score on a scale | 1.71 (0.72) | 1.83 (0.85)

29. Secondary Outcome: Student Norms Toward Violence as Assessed by the Acceptance of Dating Abuse Survey- Girls Aggressing Boys Subscale
Description: as for outcome 28
Time Frame: About 2 months after baseline
Population: Data were not collected from 1 participant in the Intervention arm because they did not answer this question. Data were not collected from 4 participants in the Control arm because they did not answer this question.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 25 | 54
score on a scale | 1.83 (0.87) | 1.67 (0.72)

30. Secondary Outcome: Student Norms Toward Violence for Girls as Assessed by the Acceptance of Dating Abuse Survey - Girls Aggressing Boy Subscale
Description: The Acceptance of Dating Abuse Survey is a questionnaire to assess among adolescents' perceptions of their norm toward violence for boys and girls. A 6-item boys aggressing girls subscale is scored as 1 (Strongly Disagree) to 4 (Strongly Agree) for each item. Then a composite score is created. The higher the number the more accepting of boys aggressing girls under certain circumstances.
Time Frame: 6 months after baseline
Population: Data were not collected from 8 participants in the Intervention arm because they did not answer this question.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 22 | 49
score on a scale | 1.70 (0.91) | 1.57 (0.67)

31. Secondary Outcome: Conflict Resolution Skills as Assessed by the Constructive Conflict Resolution Skill Subscale
Description: The Constructive and Destructive Conflict Resolution Skills questionnaire measures communication skills (Foshee et al., 2001). A 7-item constructive conflict resolution skills subscale was scored as 0 (never) to 3 (very often) for each item with a total average score ranging from 0 to 3. Higher scores reflect greater use of constructive conflict resolution skills.
Time Frame: Baseline
Population: Data were not collected from 3 participants in the Intervention arm because they did not answer this question. Data were not collected from 3 participants in the Control arm because they did not answer this question.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 40 | 77
score on a scale | 1.48 (0.92) | 1.41 (0.85)

32. Secondary Outcome: Conflict Resolution Skills as Assessed by the Constructive Conflict Resolution Skill Subscale
Description: as for outcome 31
Time Frame: about 2 months after baseline
Population: Data were not collected from 2 participants in the Intervention arm because they did not answer this question. Data were not collected from 2 participants in the Control arm because they did not answer this question.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 24 | 56
score on a scale | 1.75 (0.76) | 1.73 (0.75)

33. Secondary Outcome: Conflict Resolution Skills as Assessed by the Constructive Conflict Resolution Skill Subscale
Description: as for outcome 31
Time Frame: 6 months after baseline
Population: Data were not collected from 6 participants in the Intervention arm because they did not answer this question. Data were not collected from 1 participant in the Control arm because they did not answer this question.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 24 | 48
score on a scale | 1.35 (0.79) | 1.41 (0.78)

34. Secondary Outcome: Conflict Resolution Skills as Assessed by the Destructive Conflict Resolution Skill Subscale
Description: The Constructive and Destructive Conflict Resolution Skills questionnaire measures communication skills (Foshee et al., 2001). A 6-item destructive conflict resolution skills subscale was scored as 0 (never) to 3 (very often) for each item with a total average score ranging from 0 to 3. Higher scores reflect greater use of destructive conflict resolution skills.
Time Frame: Baseline
Population: Data were not collected from 2 participants in the Intervention arm because they did not answer this question. Data were not collected from 3 participants in the Control arm because they did not answer this question.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 41 | 77
score on a scale | 0.98 (0.83) | 0.87 (0.69)

35. Secondary Outcome: Conflict Resolution Skills as Assessed by the Destructive Conflict Resolution Skill Subscale
Description: as for outcome 34
Time Frame: about 2 months after baseline
Population: Data were not collected from 2 participants in the Intervention arm because they did not answer this question. Data were not collected from 4 participants in the Control arm because they did not answer this question.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 24 | 54
score on a scale | 1.09 (0.70) | 1.02 (0.63)

36. Secondary Outcome: Conflict Resolution Skills as Assessed by the Destructive Conflict Resolution Skill Subscale
Description: Constructive and Destructive Conflict Resolution Skills measure communication skills. A 7-item destructive conflict resolution skills subscale was scored as 0 (never) to 3 (very often) for each item. Subscale total score was created as a composite score ranging from 0 to 3 with the higher scores indicated greater use of destructive conflict resolution skills.
Time Frame: 6 months after baseline
Population: Data were not collected from 6 participants in the Intervention arm because they did not answer this question.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 24 | 49
score on a scale | 1.00 (0.70) | 0.80 (0.58)

37. Secondary Outcome: Attitudes Towards Sexting as Assessed by a One-Item Questionnaire
Description: This item assesses attitudes toward sexting among adolescents (Strassberg et al., 2013). Answer choices include: "It is always wrong to send or forward such pictures or videos" (1), "It is ok to send such pictures or videos of yourself, but not of other people" (2), "It is ok to forward such pictures or videos you might receive, but not to be the one to first send such a picture or video" (3), and "Sending, receiving, or forwarding such pictures or videos is ok" (4). Total scores range from 1-4. Higher scores reflect more positive attitudes towards sexting.
Time Frame: Baseline
Population: Data were not collected from 1 participant in the Intervention arm because they did not answer this question. Data were not collected from 3 participants in the Control arm because they did not answer this question
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 42 | 77
score on a scale | 1.26 (0.63) | 1.345 (0.85)

38. Secondary Outcome: Attitudes Towards Sexting as Assessed by a One-Item Questionnaire
Description: as for outcome 37
Time Frame: about 2 months after intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 26 | 58
score on a scale | 1.42 (0.70) | 1.41 (0.84)

39. Secondary Outcome: Attitudes Towards Sexting as Assessed by a One-Item Questionnaire
Description: as for outcome 37
Time Frame: 6 months after intervention
Population: Data were not collected from 4 participants in the Intervention arm because they did not answer this question.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 26 | 49
score on a scale | 1.15 (0.46) | 1.37 (0.86)

40. Secondary Outcome: Perceived Parental Communication About Different Topics as Assessed by One-Item From an Adapted Version of the Modified Miller Communication Scale
Description: This item assesses perceived parental communication about different topics (how to handle problems in relationships, how to handle emotions, appropriate behavior when communicating through technology [texting/social networking], what's important to you and/or parent/caregiver [values] when it comes to romantic relationships, choosing your dating partners, none of the above) adapted from the Modified Miller Communication Scale (Rizzo et al., 2001; Miller et al., 1998). Scores reflect the number of topics discussed by the parent/guardian and child. The higher the number, the more topics discussed.
Time Frame: Baseline
Population: One intervention arm participant and three control arm participants provided inconsistent responses by indicating they talked about at least one topic and also reported not discussing these topics with their parent/caregiver. These inconsistent responses were set to missing.
Measure: Mean (Standard Deviation); unit: number of topics
Arm/Group | Intervention | Control
Number analyzed (Participants) | 42 | 77
number of topics | 1.21 (1.37) | 1.21 (1.21)

41. Secondary Outcome: Perceived Parental Communication About Different Topics as Assessed by One-Item From an Adapted Version of the Modified Miller Communication Scale
Description: as for outcome 40
Time Frame: about 2 months after Baseline
Population: 2 control arm participants provided inconsistent responses by indicating they talked about at least one topic and also reported not discussing these topics with their parent/caregiver. These inconsistent responses were set to missing.
Measure: Mean (Standard Deviation); unit: number of topics
Arm/Group | Intervention | Control
Number analyzed (Participants) | 26 | 56
number of topics | 1.12 (1.07) | 1.79 (1.44)

42. Secondary Outcome: Perceived Parental Communication About Different Topics as Assessed by One-Item From an Adapted Version of the Modified Miller Communication Scale
Description: as for outcome 40
Time Frame: 6 months after Baseline
Measure: Mean (Standard Deviation); unit: number of topics
Arm/Group | Intervention | Control
Number analyzed (Participants) | 30 | 49
number of topics | 0.73 (0.98) | 1.78 (1.75)

43. Secondary Outcome: Perceived Frequency of Parental Communication About Different Topics as Assessed by One-Item From an Adapted Version of the Modified Miller Communication Scale
Description: This item assesses perceived frequency of parental communication about different topics adapted from the Modified Miller Communication Scale (Rizzo et al., 2001; Miller et al., 1998). It is scored from 1 (never) to 4 (a lot; more than 3 times) with total scores ranging from 1-4. Higher scores reflect greater frequency of communication about topics.
Time Frame: Baseline
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 42 | 78
score on a scale | 1.98 (1.18) | 1.83 (0.99)

44. Secondary Outcome: Perceived Frequency of Parental Communication About Different Topics as Assessed by One-Item From an Adapted Version of the Modified Miller Communication Scale
Description: as for outcome 43
Time Frame: about 2 months after baseline
Population: Data were not collected from 1 participant in the Intervention arm because they did not answer this question. Data were not collected from 1 participant in the Control arm because they did not answer this question .
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 25 | 57
score on a scale | 1.84 (1.07) | 2.05 (1.01)

45. Secondary Outcome: Perceived Frequency of Parental Communication About Different Topics as Assessed by One-Item From an Adapted Version of the Modified Miller Communication Scale
Description: as for outcome 43
Time Frame: 6 months after baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 30 | 49
score on a scale | 1.73 (0.94) | 1.82 (0.97)

46. Secondary Outcome: Perceived Helpfulness of Parental Communication About Different Topics as Assessed by One-Item From an Adapted Version of the Modified Miller Communication Scale
Description: This item assesses perceived helpfulness of communication about different topics with parents/guardians adapted from the Modified Miller Communication Scale (Rizzo et al., 2001; Miller et al., 1998). It is scored from 1 (not at all helpful) to 7 (very helpful) with total scores ranging from 1-7. Higher scores reflect greater perceived helpfulness of communication about topics.
Time Frame: Baseline
Population: Data were not collected from 17 participants in the Intervention arm because they did not answer this question. Data were not collected from 29 participants in the Control arm because they did not answer this question.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 26 | 51
score on a scale | 4.31 (2.24) | 4.55 (1.90)

47. Secondary Outcome: Perceived Helpfulness of Parental Communication About Different Topics as Assessed by One-Item From an Adapted Version of the Modified Miller Communication Scale
Description: as for outcome 46
Time Frame: about 2 months after baseline
Population: Data were not collected from 10 participants in the Intervention arm because they did not answer this question. Data were not collected from 17 participants in the Control arm because they did not answer this question
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 16 | 41
score on a scale | 4.25 (1.95) | 4.20 (1.81)

48. Secondary Outcome: Perceived Helpfulness of Parental Communication About Different Topics as Assessed by One-Item From an Adapted Version of the Modified Miller Communication Scale
Description: as for outcome 46
Time Frame: 6 months after baseline
Population: Data were not collected from 16 participants in the Intervention arm because they did not answer this question. Data were not collected from 18 participants in the Control arm because they did not answer this question.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 14 | 31
score on a scale | 4.43 (2.10) | 4.42 (1.91)

49. Secondary Outcome: Perceived Comfort of Parental Communication About Different Topics as Assessed by One-Item From an Adapted Version of the Modified Miller Communication Scale
Description: This item assesses perceived comfort of communication about different topics with parents/guardians adapted from the Modified Miller Communication Scale (Rizzo et al., 2001; Miller et al., 1998). It is scored from 1 (not at all comfortable) to 7 (very comfortable) with total scores ranging from 1-7. Higher scores reflect greater perceived comfort in communicating with parents/guardians about topics.
Time Frame: Baseline
Population: Data were not collected from 17 participants in the Intervention arm because they did not answer this question. Data were not collected from 31 participants in the Control arm because they did not answer this question.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 26 | 49
score on a scale | 4.12 (1.97) | 4.27 (1.86)

50. Secondary Outcome: Perceived Comfort of Parental Communication About Different Topics as Assessed by One-Item From an Adapted Version of the Modified Miller Communication Scale
Description: as for outcome 49
Time Frame: about 2 months after baseline
Population: Data were not collected from 10 participants in the Intervention arm because they did not answer this question. Data were not collected from 19 participants in the Control arm because they did not answer this question
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 16 | 39
score on a scale | 4.81 (2.01) | 3.87 (1.69)

51. Secondary Outcome: Perceived Comfort of Parental Communication About Different Topics as Assessed by One-Item From an Adapted Version of the Modified Miller Communication Scale
Description: as for outcome 49
Time Frame: 6 months after baseline
Population: as for outcome 48
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 14 | 31
score on a scale | 4.21 (1.97) | 4.32 (1.87)

52. Secondary Outcome: Perceived Parental Comfort of Parental Communication About Different Topics as Assessed by One-Item From an Adapted Version of the Modified Miller Communication Scale
Description: This item assesses perceived parental comfort of parental communication about different topics adapted from the Modified Miller Communication Scale (Rizzo et al., 2001; Miller et al., 1998). It is scored from 1 (not at all comfortable) to 7 (very comfortable) with total scores ranging from 1-7. Higher scores reflect greater perceived parental comfort in communicating about topics.
Time Frame: Baseline
Population: Data were not collected from 17 participants in the Intervention arm because they did not answer this question. Data were not collected from 30 participants in the Control arm because they did not answer this question.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 26 | 50
score on a scale | 4.81 (1.79) | 4.84 (1.97)

53. Secondary Outcome: Perceived Parental Comfort of Parental Communication About Different Topics as Assessed by One-Item From an Adapted Version of the Modified Miller Communication Scale
Description: as for outcome 52
Time Frame: about 2 months after baseline
Population: Data were not collected from 10 participants in the Intervention arm because they did not answer this question. Data were not collected from 18 participants in the Control arm because they did not answer this question.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 16 | 40
score on a scale | 4.88 (2.00) | 4.33 (1.94)

54. Secondary Outcome: Perceived Parental Comfort of Parental Communication About Different Topics as Assessed by One-Item From an Adapted Version of the Modified Miller Communication Scale
Description: as for outcome 52
Time Frame: 6 months after baseline
Population: Data were not collected from 16 participants in the Intervention arm because they did not answer this question. Data were not collected from 20 participants in the Control arm because they did not answer this question.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 14 | 29
score on a scale | 4.29 (1.91) | 4.34 (1.88)

55. Secondary Outcome: Perceived Confidence in Communication About Different Topics With Parent as Assessed by a One-Item Questionnaire
Description: This item assesses perceived confidence in communicating about different topics with parents/guardian (Foshee et al., 2012). It is scored from 1 (very confident) to 4 (not at all confident) total mean scores ranging from 1-4. Higher scores reflect lower perceived confidence in communicating about topics with parents/guardians.
Time Frame: Baseline
Population: as for outcome 49
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 26 | 49
score on a scale | 1.88 (0.82) | 2.33 (1.01)

56. Secondary Outcome: Perceived Confidence in Communication About Different Topics With Parent as Assessed by a One-Item Questionnaire
Description: as for outcome 55
Time Frame: about 2 months after baseline
Population: as for outcome 53
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 16 | 40
score on a scale | 2.13 (1.15) | 2.10 (0.96)

57. Secondary Outcome: Perceived Confidence in Communication About Different Topics With Parent as Assessed by a One-Item Questionnaire
Description: as for outcome 55
Time Frame: 6 months after baseline
Population: as for outcome 48
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 14 | 31
score on a scale | 1.79 (0.89) | 2.16 (0.90)

58. Secondary Outcome: Youth's Attitudes Towards Need for Consent as Assessed by the Adapted Version of the Sexual Consent Scale-Revised
Description: An adapted 8-item version of the sexual consent- scale revised was used to assess youth attitudes towards need for consent (Humphreys et al., 2010). Each item was scored from 1 (Strongly Disagree) to 4 (Strongly Agree) and an average score was calculated, ranging from 1-4. Higher scores reflect more positives attitudes toward need for consent.
Time Frame: Baseline
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 40 | 74
score on a scale | 3.11 (0.66) | 2.894 (0.86)

59. Secondary Outcome: Youth's Attitudes Towards Need for Consent as Assessed by the Adapted Version of the Sexual Consent Scale-Revised
Description: as for outcome 58
Time Frame: about 2 months after baseline
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 23 | 52
score on a scale | 3.23 (0.66) | 2.96 (0.81)

60. Secondary Outcome: Youth's Attitudes Towards Need for Consent as Assessed by the Adapted Version of the Sexual Consent Scale-Revised
Description: as for outcome 58
Time Frame: 6 months after baseline
Population: Data were not collected from 5 participants in the Intervention arm because they did not answer this question. Data were not collected from 2 participants in the Control arm because they did not answer this question.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 25 | 47
score on a scale | 3.10 (0.73) | 2.96 (0.69)

61. Secondary Outcome: Knowledge of the Select, Detect, Protect Decision-Making Paradigm as Assessed by a One-Item Questionnaire
Description: This item assesses knowledge of the "select, detect, protect" decision-making paradigm (a core feature in the curriculum). Respondents choose from five possible responses that include different combinations of the paradigm, with one response being the correct answer. The item is scored as 0 (not correct) or 1 (correct). Results are reported as the number of respondents who selected the correct response and the number who selected an incorrect response.
Time Frame: Baseline
Population: Data were not collected from 2 participants in the Control arm because they did not answer this question.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 43 | 78
Participants
  Correct | 3 | 15
  Incorrect | 40 | 63

62. Secondary Outcome: Knowledge of the Select, Detect, Protect Decision-Making Paradigm as Assessed by a One-Item Questionnaire
Description: as for outcome 61
Time Frame: about 2 months after baseline
Population: Data were not collected from 1 participant in the Control arm because they did not answer this question.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 26 | 57
Participants
  Correct | 10 | 13
  Incorrect | 16 | 44

63. Secondary Outcome: Knowledge of the Select, Detect, Protect Decision-Making Paradigm as Assessed by a One-Item Questionnaire
Description: as for outcome 61
Time Frame: 6 months after baseline
Population: Data were not collected from 4 participants in the Intervention arm because they did not answer this question. Data were not collected from 2 participants in the Control arm because they did not answer this question.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 26 | 47
Participants
  Correct | 7 | 5
  Incorrect | 19 | 42

64. Secondary Outcome: Responsible Decision-Making as Assessed by the Social and Emotional Competency Assessment - The Responsible Decision-Making Subscale
Description: The Washoe County School District (WCSD) Social and Emotional Competency Assessment (Short Form) includes 17 items, including a 4-item Responsible Decision-Making subscale that assesses how easy or difficult it is to make responsible decisions. It is scored from 1 (Very Difficult) to 4 (Very Easy) for each item with a total average score ranging from 1-4. Higher scores reflect a greater ability to make responsible decisions.
Time Frame: Baseline
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 42 | 76
score on a scale | 2.91 (0.65) | 2.78 (0.79)

65. Secondary Outcome: Responsible Decision-Making as Assessed by the Social and Emotional Competency Assessment - The Responsible Decision-Making Subscale
Description: as for outcome 64
Time Frame: about 2 months after baseline
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 24 | 56
score on a scale | 2.95 (0.59) | 2.65 (0.67)

66. Secondary Outcome: Responsible Decision-Making as Assessed by the Social and Emotional Competency Assessment - The Responsible Decision-Making Subscale
Description: as for outcome 64
Time Frame: 6 months after baseline
Population: Data were not collected from 6 participants in the Intervention arm because they did not answer this question. Data were not collected from 3 participants in the Control arm because they did not answer this question.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 24 | 46
score on a scale | 2.81 (0.67) | 2.70 (0.75)

67. Secondary Outcome: Emotional Regulation as Assessed by the Social and Emotional Competency Assessment - The Emotional Regulation Subscale
Description: The Washoe County School District (WCSD) Social and Emotional Competency Assessment (Short Form) includes 17 items, including a 4-item Emotional Regulation subscale that assesses how easy or difficult it is to use emotional regulation skills. It is scored from 1 (Very Difficult) to 4 (Very Easy) for each item with a total average score ranging from 1-4. Higher scores reflect a greater ability to use emotional regulation skills.
Time Frame: Baseline
Population: Data were not collected from 4 participants in the Control arm because they did not answer this question.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 43 | 76
score on a scale | 2.52 (0.80) | 2.40 (0.82)

68. Secondary Outcome: Emotional Regulation as Assessed by the Social and Emotional Competency Assessment - The Emotional Regulation Subscale
Description: as for outcome 67
Time Frame: about 2 months after baseline
Population: Data were not collected from 2 participants in the Intervention arm because they did not answer this question. Data were not collected from 1 participant in the Control arm because they did not answer this question.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 24 | 57
score on a scale | 2.43 (0.72) | 2.33 (0.72)

69. Secondary Outcome: Emotional Regulation as Assessed by the Social and Emotional Competency Assessment - The Emotional Regulation Subscale
Description: as for outcome 67
Time Frame: 6 months after baseline
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 24 | 48
score on a scale | 2.35 (0.78) | 2.43 (0.79)

70. Secondary Outcome: Youth's Goal Management as Assessed by the Social and Emotional Competency Assessment - Goal Management Subscale
Description: The Washoe County School District (WCSD) Social and Emotional Competency Assessment (Short Form) includes 17 items, including a 4-item Goal Management subscale that assesses how easy or difficult it is to manage goals. It is scored from 1 (Very Difficult) to 4 (Very Easy) for each item with a total average score ranging from 1-4. Higher scores reflect a greater ability to manage goals
Time Frame: Baseline
Population: Data were not collected from 2 participants in the Intervention arm because they did not answer this question. Data were not collected from 5 participants in the Control arm because they did not answer this question.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 41 | 75
score on a scale | 2.73 (0.79) | 2.52 (0.87)

71. Secondary Outcome: Youth's Goal Management as Assessed by the Social and Emotional Competency Assessment - Goal Management Subscale
Description: as for outcome 70
Time Frame: about 2 months after baseline
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 24 | 55
score on a scale | 2.74 (0.74) | 2.50 (0.66)

72. Secondary Outcome: Youth's Goal Management as Assessed by the Social and Emotional Competency Assessment - Goal Management Subscale
Description: as for outcome 70
Time Frame: 6 months after baseline
Population: Data were not collected from 4 participants in the Intervention arm because they did not answer this question. Data were not collected from 3 participants in the Control arm because they did not answer this question
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 26 | 46
score on a scale | 2.67 (0.95) | 2.63 (0.76)

73. Secondary Outcome: Youth's Emotional Knowledge as Assessed by the Social and Emotional Competency Assessment - Emotional Knowledge Subscale
Description: The Washoe County School District (WCSD) Social and Emotional Competency Assessment (Short Form) includes 17 items, including a 2-item Emotional Knowledge subscale that assesses how easy or difficult it is to use emotional knowledge. It is scored from 1 (Very Difficult) to 4 (Very Easy) for each item with a total average score ranging from 1-4. Higher scores reflect a greater ability to use emotional knowledge.
Time Frame: Baseline
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 41 | 77
score on a scale | 2.79 (0.82) | 2.62 (0.92)

74. Secondary Outcome: Youth's Emotional Knowledge as Assessed by the Social and Emotional Competency Assessment - Emotional Knowledge Subscale
Description: as for outcome 73
Time Frame: about 2 months after baseline
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 24 | 55
score on a scale | 2.94 (0.77) | 2.65 (0.76)

75. Secondary Outcome: Youth's Emotional Knowledge as Assessed by the Social and Emotional Competency Assessment - Emotional Knowledge Subscale
Description: as for outcome 73
Time Frame: 6 months after baseline
Population: Data were not collected from 4 participants in the Intervention arm because they did not answer this question. Data were not collected from 1 participant in the Control arm because they did not answer this question.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 26 | 48
score on a scale | 2.65 (0.87) | 2.61 (0.81)

76. Secondary Outcome: Youth's Likeliness to Seek Help From a Parent/Caregiver as Assessed by One Item From the General Help-Seeking Questionnaire
Description: One item assessing youth's likeliness to seek help from a parent/caregiver if they were having a problem with relationships was adapted from the General Help-Seeking Questionnaire (Wilson et al., 2005). The item is scored from 1 (very unlikely to seek support) to 4 (very likely to seek support) with total scores ranging from 1 to 4. Higher scores reflect greater likeliness to seek help.
Time Frame: Baseline
Population: Data were not collected from 2 participants in the Intervention arm because they did not answer this question. Data were not collected from 6 participants in the Control arm because they did not answer this question.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 41 | 74
score on a scale | 2.54 (1.14) | 2.51 (1.28)

77. Secondary Outcome: Youth's Likeliness to Seek Help From a Parent/Caregiver as Assessed by One Item From the General Help-Seeking Questionnaire
Description: as for outcome 76
Time Frame: about 2 months after baseline
Population: Data were not collected from 2 participants in the Control arm because they did not answer this question.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 26 | 56
score on a scale | 2.73 (1.08) | 2.70 (1.09)

78. Secondary Outcome: Youth's Likeliness to Seek Help From a Parent/Caregiver as Assessed by One Item From the General Help-Seeking Questionnaire
Description: as for outcome 76
Time Frame: 6 months after baseline
Population: as for outcome 60
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 25 | 47
score on a scale | 2.68 (1.14) | 2.77 (1.05)

79. Secondary Outcome: Bullying Perpetration as Assessed by Adapted Olweus Bully/Victim Questionnaire for Students - Bully Perpetration Subscale
Description: The adapted Olweus Bully/Victim Questionnaire for Students includes 16 items with an 8-item Bully Perpetration subscale (Olweus, 1996). Response options for each item include: 0 (Never), 1 (rarely), 2 (Occasionally), 3 (somewhat often), 4 (Often). Perpetrators are counted as those youth who respond with options 2, 3, or 4 to any item.
Time Frame: Baseline
Population: as for outcome 26
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 42 | 78
Participants
  "Yes" Considered Perpetrators | 11 | 21
  "No" Not Considered Perpetrators | 31 | 57

80. Secondary Outcome: Bullying Perpetration as Assessed by Adapted Olweus Bully/Victim Questionnaire for Students - Bully Perpetration Subscale
Description: as for outcome 79
Time Frame: 6 months after baseline
Population: Data were not collected from 3 participants in the Intervention arm because they did not answer this question. Data were not collected from 1 participant in the Control arm because they did not answer this question.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 27 | 48
Participants
  "Yes" Considered Perpetrators | 5 | 7
  "No" Not Considered Perpetrators | 22 | 41

81. Secondary Outcome: Bully Victimization as Assessed by Adapted Olweus Bully/Victim Questionnaire for Students - Bully Victimization Subscale
Description: The adapted Olweus Bully/Victim Questionnaire for Students includes 16 items with an 8-item Bully Victimization subscale (Olweus, 1996). Response options for each item include: 0 (Never), 1 (rarely), 2 (Occasionally), 3 (somewhat often), 4 (Often). Victims are counted as those youth who respond with options 2, 3, or 4 to any item.
Time Frame: Baseline
Population: Data were not collected from 2 participants in the Control arm because they did not answer this question.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 43 | 78
Participants
  "Yes" Considered Victims | 18 | 33
  "No" Not Considered Victims | 25 | 45

82. Secondary Outcome: Bully Victimization as Assessed by Adapted Olweus Bully/Victim Questionnaire for Students - Bully Victimization Subscale
Description: as for outcome 81
Time Frame: 6 months after baseline
Population: Data were not collected from 3 participants in the Intervention arm because they did not answer this question.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 27 | 49
Participants
  "Yes" Considered Victims | 10 | 19
  "No" Not Considered Victims | 17 | 30

83. Secondary Outcome: Youth's Perception of Caregiver Communication as Assessed by a One-Item Questionnaire
Description: This one item assesses youth's perception of the frequency with which their caregiver engaged in critical communication with them during the past month (adapted from Foshee et al., 2012). The item was scored as 0 (none of the time) to 4 (all of the time) with higher scores indicating a higher frequency of critical communication.
Time Frame: Baseline
Population: Data were not collected from 3 participants in the Control arm because they did not answer this question.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 43 | 77
score on a scale | 1.35 (1.29) | 1.62 (1.50)

84. Secondary Outcome: Youth's Perception of Caregiver Communication as Assessed by a One-Item Questionnaire
Description: as for outcome 83
Time Frame: 6 months after baseline
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 25 | 48
score on a scale | 1.60 (1.61) | 1.56 (1.38)

85. Secondary Outcome: Youth Perception of Caregiver Rules About Dating as Assessed by a Questionnaire
Description: This 7-item scale assesses youth's perception of the number of caregiver's rules about dating (Foshee et al., 2012). Responses include yes and no for each item; for four of the items, there was also a 'don't know' option. Total average score ranges from 0 to 7, with higher scores reflecting greater perceptions of the number (or count) of rules their caregiver has about dating.
Time Frame: Baseline
Population: Data were not collected from 1 participant in the Intervention arm because they did not answer this question. Data were not collected from 11 participants in the Control arm because they did not answer this question.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 42 | 69
score on a scale | 3.79 (2.45) | 3.41 (2.38)

86. Secondary Outcome: Youth Perception of Caregiver Rules About Dating as Assessed by a Questionnaire
Description: as for outcome 85
Time Frame: 6 months after baseline
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 24 | 48
score on a scale | 3.88 (2.61) | 3.46 (2.67)

87. Secondary Outcome: Youth Perception of Parental Monitoring as Assessed by a Questionnaire
Description: This 5-item scale assesses youth's perception of how much their parents or caregivers know about what the youth is doing with regards to their friends, how they spend their money, etc. (Brown et al., 1993). The items were scored as 1 (don't know much) to 4 (know a lot) with a total average score ranging from 1 to 4. Higher scores reflect greater perceptions of parental monitoring.
Time Frame: Baseline
Population: Data were not collected from 6 participants in the Intervention arm because they did not answer this question. Data were not collected from 9 participants in the Control arm because they did not answer this question.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 37 | 71
score on a scale | 2.97 (0.79) | 2.79 (0.93)

88. Secondary Outcome: Youth Perception of Parental Monitoring as Assessed by a Questionnaire
Description: as for outcome 87
Time Frame: 6 months after baseline
Population: as for outcome 60
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 25 | 47
score on a scale | 2.80 (1.06) | 2.90 (0.89)

89. Secondary Outcome: Youth Perceived Parental Closeness as Assessed by a Questionnaire
Description: This 6-item scale assesses youth's perception of their perceived closeness with their parent/caregiver (Vazsonyi et al., 2003). It is scored from 1 (strongly disagree) to 5 (strongly agree) for each item with an average score ranging from 1 to 5. Higher scores reflect greater parental closeness.
Time Frame: Baseline
Population: Data were not collected from 3 participants in the Intervention arm because they did not answer this question. Data were not collected from 9 participants in the Control arm because they did not answer this question.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 40 | 71
score on a scale | 3.59 (1.10) | 3.45 (1.19)

90. Secondary Outcome: Youth Perceived Parental Closeness as Assessed by a Questionnaire
Description: as for outcome 89
Time Frame: 6 months after baseline
Population: Data were not collected from 7 participants in the Intervention arm because they did not answer this question. Data were not collected from 1 participant in the Control arm because they did not answer this question.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 23 | 48
score on a scale | 3.57 (1.03) | 3.39 (1.01)

91. Secondary Outcome: Youth's Perception of Their School Climate as Assessed by Survey Items From the Dating Matters School Educator Survey
Description: This 4-item scale, adapted from items in the Dating Matters School Educator Survey, assesses youth perception of the general school climate (Niolon et al., 2019). Each item is scored from 1 (strongly disagree) to 5 (strongly agree) with a total average score ranging from 1-5. Higher scores reflect more positive perceptions of school climate.
Time Frame: Baseline
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 40 | 74
score on a scale | 3.28 (0.96) | 3.33 (1.10)

92. Secondary Outcome: Youth's Perception of Their School Climate as Assessed by Survey Items From the Dating Matters School Educator Survey
Description: as for outcome 91
Time Frame: 6 months after baseline
Population: as for outcome 66
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 24 | 46
score on a scale | 3.40 (0.96) | 3.10 (0.97)

93. Secondary Outcome: Youth's Perception of Their School's Teen Dating Violence Climate as Assessed by Survey Items From the Dating Matters School Educator Survey
Description: This 6-item scale, adapted from items in the Dating Matters School Educator Survey, assesses the perceived frequency with which certain behaviors are observed among students who are dating in the school. This was scored from 0 (Never) to 3 (Often) with a total average score ranging from 0-3. Higher scores reflect greater perceived frequency of observing the behaviors.
Time Frame: Baseline
Population: Data were not collected from 5 participants in the Intervention arm because they did not answer this question. Data were not collected from 9 participants in the Control arm because they did not answer this question.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 38 | 71
score on a scale | 0.51 (0.68) | 0.38 (0.68)

94. Secondary Outcome: Youth's Perception of Their School's Teen Dating Violence Climate as Assesed by Survey Items From the Dating Matters School Educator Survey
Description: as for outcome 93
Time Frame: 6 months after baseline
Population: as for outcome 66
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 24 | 46
score on a scale | 0.53 (0.74) | 0.66 (0.85)

95. Secondary Outcome: Knowledge of Human Trafficking as Assessed by a Questionnaire
Description: A 5-item questionnaire, adapted from the U.S. Department of Homeland Security 'Blue Campaign', was used to asses youth knowledge of human trafficking. Youth are presented with 5 items which they have to designate as 'true' or 'false" about human trafficking. Each item is scored as 1 (correct) or 0 (incorrect). Total score is computed as the percent of items answered correctly which translates into a mean score ranging from 0-1, with higher score indicating greater knowledge.
Time Frame: Baseline
Population: Data were not collected from 2 participants in the Intervention arm because they did not answer this question. Data were not collected from 7 participants in the Control arm because they did not answer this question.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 41 | 73
score on a scale | 0.45 (0.29) | 0.53 (0.32)

96. Secondary Outcome: Knowledge of Human Trafficking as Assessed by a Questionnaire
Description: as for outcome 95
Time Frame: about 2 months after baseline
Population: Data were not collected from 1 participant in the Intervention arm because they have were lost to follow up. Data were not collected from 3 participants in the Control arm because they were lost of follow up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 25 | 55
score on a scale | 0.37 (0.20) | 0.44 (0.28)

97. Secondary Outcome: Knowledge of Human Trafficking as Assessed by a Questionnaire
Description: as for outcome 95
Time Frame: 6 months after baseline
Population: Data were not collected from 5 participants in the Intervention arm because they have were lost to follow up. Data were not collected from 1 participant in the Control arm because they were lost of follow up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 25 | 48
score on a scale | 0.55 (0.28) | 0.46 (0.29)

98. Secondary Outcome: Perception of Positive Relationship Skills as Assessed by a Questionnaire
Description: This 4-item questionnaire assesses youth perception of the frequency with which their most recent dating partner engaged in positive relationship skills with them (Niolon et al., 2019). The items are scored from 0 (Never) to 3 (Always) with a total average score ranging from 0 to 3. Higher scores reflect greater perceived frequency of more positive relationship skills.
Time Frame: Baseline
Population: Data were not collected from 27 participants in the Intervention arm because they did not answer this question. Data were not collected from 52 participants in the Control arm because they did not answer this question.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 16 | 28
score on a scale | 2.11 (0.94) | 1.84 (0.94)

99. Secondary Outcome: Perception of Positive Relationship Skills as Assessed by a Questionnaire
Description: as for outcome 98
Time Frame: 6 months after baseline
Population: Data were not collected from 24 participants in the Intervention arm because they did not answer this question. Data were not collected from 33 participants in the Control arm because they did not answer this question.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 6 | 16
score on a scale | 1.79 (1.12) | 1.88 (0.85)

100. Secondary Outcome: Perception of Peer Risk Behaviors as Assessed by the Perception of Peer In-Person and Electronic Dating Violence Perpetration Subscale
Description: The Perception of Peer Risk Behaviors measure includes 7 items, including a 4-item 'Perception of Peer In-Person and Electronic Dating Violence Perpetration' subscale, that assesses youth perception of the total number of friends who engage in in-person or electronic dating violence perpetration. It is scored from 1 (None of them) to 5 (All of them) for each item with a total average score ranging from 1 to 5. Higher scores reflect greater perception of peer in-person and electronic dating violence perpetration.
Time Frame: Baseline
Population: Data were not collected from 1 participant in the Intervention arm because they did not answer this question. Data were not collected from 5 participants in the Control arm because they did not answer this question.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 42 | 75
score on a scale | 1.20 (0.42) | 1.29 (0.91)

101. Secondary Outcome: Perception of Peer Risk Behaviors as Assessed by the Perception of Peer In-Person and Electronic Dating Violence Perpetration Subscale
Description: as for outcome 100
Time Frame: 6 months after baseline
Population: Data were not collected from 5 participants in the Intervention arm because they did not answer this question.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 25 | 49
score on a scale | 1.18 (0.58) | 1.10 (0.47)

102. Secondary Outcome: Perception of Peer Risk Behaviors as Assessed by the Perception of Peer Substance Use and Fighting Subscale
Description: The Perception of Peer Risk Behaviors measure includes 7 items, including a 3-item 'Perception of Peer Substance Use and Fighting' subscale, that assesses youth perception of the total number of friends who engage in substance use and fighting. It is scored from 1 (None of them) to 5 (All of them) for each item with a total average score ranging from 1 to 5. Higher scores reflect greater perception of peer substance use and fighting.
Time Frame: Baseline
Population: as for outcome 95
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 41 | 73
score on a scale | 1.58 (0.73) | 1.71 (0.96)

103. Secondary Outcome: Perception of Peer Risk Behaviors as Assessed by the Perception of Peer Substance Use and Fighting Subscale
Description: as for outcome 102
Time Frame: 6 months after baseline
Population: Data were not collected from 4 participants in the Intervention arm because they did not answer this question.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 26 | 49
score on a scale | 1.33 (0.52) | 1.50 (0.69)

ADVERSE EVENTS:
Time Frame: Up to 6 months
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/80
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/80
Other Adverse Events (participants affected / at risk) | 0/43 | 0/80

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2023-12-08): https://cdn.clinicaltrials.gov/large-docs/27/NCT05225727/Prot_000.pdf
  • Informed Consent Form (2022-09-16): https://cdn.clinicaltrials.gov/large-docs/27/NCT05225727/ICF_001.pdf